CLINICAL TRIAL: NCT07392307
Title: Association Between Dry Eye Disease and Diabetic Macular Edema
Acronym: DED-DME
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Aly, Resident doctor, Ophthalmology department, sohag teaching hospital, Sohag University
Other Study IDs: EAly
Record Dates: First submitted 2026-01-27; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Disease (DED) , Diabetic Macular Edema
Keywords: Dry eye disease; Diabetic macular edema; Diabetes mellitus; Ocular surface; Optical coherence tomography (OCT); Ophthalmology
MeSH Terms: conditions — Dry Eye Syndromes; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Participants with Diabetic Macular Edema (DME): Participants diagnosed with DME. Dry Eye Disease (DED) will be assessed using imaging and clinical evaluation (OSDI questionnaire, TBUT, Schirmer test, ocular surface examination).
  Interventions: Diagnostic Test: Dry Eye Disease Assessment
- Group 2: Participants without DME: Participants without DME. Dry Eye Disease (DED) will be assessed using imaging and clinical evaluation (OSDI questionnaire, TBUT, Schirmer test, ocular surface examination).
  Interventions: Diagnostic Test: Dry Eye Disease Assessment

INTERVENTIONS:
Diagnostic Test: Dry Eye Disease Assessment — Assessment of dry eye symptoms, tear film function, and ocular surface examination using standardized questionnaires and clinical tests (OSDI, TBUT, Schirmer test).

SUMMARY:
This study evaluates the association between dry eye disease (DED) and diabetic macular edema (DME) in adult patients at the Ophthalmology Department, Faculty of Medicine, Sohag University. Participants will undergo standardized assessments for dry eye and clinical evaluation for macular edema. The goal is to improve understanding of the relationship between these two eye conditions in patients with diabetes.

DETAILED DESCRIPTION:
This prospective observational cross-sectional study investigates the relationship between Dry Eye Disease (DED) and Diabetic Macular Edema (DME) in adult diabetic patients at the Ophthalmology Department, Faculty of Medicine, Sohag University.

Participants undergo comprehensive ocular assessments during a single baseline visit, including:

DED evaluation: Ocular Surface Disease Index (OSDI) questionnaire, tear film break-up time (TBUT), Schirmer test, and slit-lamp ocular surface examination.

DME assessment: Clinical fundus examination and Optical Coherence Tomography (OCT) imaging.

The study aims to identify associations between anterior segment (ocular surface) parameters and posterior segment pathology (macular edema), to improve understanding of diabetic ocular complications and inform future screening and management strategies.

The study design is cross-sectional (all assessments at a single visit) and prospective regarding enrollment and data collection at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years.
* Confirmed diagnosis of diabetes mellitus >8 years.
* Ability to undergo OCT examination.
* Ability to perform standardized dry eye diagnostic tests.
* Signed informed consent after explanation of study purpose.

Exclusion Criteria:

* History of ocular surgery.
* History of Argon laser photocoagulation.
* Advanced proliferative diabetic retinopathy (PDR): tractional retinal detachment, vitreous hemorrhage, optic neuropathy.
* Previous significant ocular trauma.
* Presence of other ocular surface diseases, or history of systemic or ocular surgeries affecting the eye.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 50 patients with diabetes aged 18-60 years, including 25 patients with diabetic macular edema and 25 patients without macular edema.
  Design : This cross-sectional observational study aims to assess ocular and systemic characteristics associated with diabetic macular edema
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Dry Eye Disease (DED) Symptom Severity | Baseline (single visit)
  DED symptoms will be assessed using the Ocular Surface Disease Index (OSDI) questionnaire to quantify ocular discomfort, visual disturbance, and functional limitations.
  Units of Measure: OSDI score (0-100)
Tear Film Function | Baseline (single visit)
  Tear film function will be evaluated using Tear Break-Up Time (TBUT) to measure tear film stability and the Schirmer test to assess tear production. Three consecutive measurements are averaged for TBUT; Schirmer test is performed over 5 minutes.
  Units of Measure: TBUT in seconds; Schirmer test in millimeters (mm)
Diabetic Macular Edema (DME) Severity | Baseline (single visit)
  Diabetic Macular Edema (DME) Severity Description: DME severity will be assessed by clinical fundus examination and Optical Coherence Tomography (OCT) imaging to determine the presence and severity of macular edema. Central macular thickness and retinal fluid are measured.
  Units of Measure: Macular thickness in micrometers (µm); clinical grading of edema.

CONTACTS AND LOCATIONS:
Overall Officials: Islam A Ahmed, MD,PhD, Study Director — Sohag University, Faculty of Medicine
Locations (1):
- Sohag university, Sohag, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Plans to share Individual Participant Data (IPD) are currently undecided. Any future sharing will follow ethical approvals, institutional policies, and measures to protect participant confidentiality.

REFERENCES:
- [Background] Manaviat MR, Rashidi M, Afkhami-Ardekani M, Shoja MR. Prevalence of dry eye syndrome and diabetic retinopathy in type 2 diabetic patients. BMC Ophthalmology. 2008;8:10.
- [Background] Craig JP, Nichols KK, Akpek EK, et al. TFOS DEWS II Definition and Classification Report. The Ocular Surface. 2017;15(3):276-283.